CLINICAL TRIAL: NCT07293338
Title: Prognostic Values of Coronary Microvascular Dysfunction in Patients With Dilated Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0971
Record Dates: First submitted 2025-11-18; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Dilated Cardiomyopathy (DCM)
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Coronary microvascular dysfunction
  Interventions: Procedure: coronary angiography
- Non-Coronary microvascular dysfunction
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: coronary angiography — Patients should undergo coronary angiography to confirm the absence of significant coronary stenosis. Angio-IMR was calculated based on the angiography.

SUMMARY:
The goal of this observational study is to learn about the long-term prognostic of coronary microvascular dysfuction in Patients with Dilated Cardiomyopathy.

The main question it aims to answer is: Does the coronary microvascular dysfunction impact the outcomes in Patients with Dilated Cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy comfirmed by echocardiography: LVDd > 55 mm in men or > 50 mm in women.
* Clinically evident congestive heart failure: Compatible symptoms and signs, and BNP ≥ 35 pg/mL or NT-proBNP ≥ 125 pg/mL, and LV systolic dysfunction defined by LVEF < 45 %.
* Coronary angiography showing stenosis ≤ 50 % in all major epicardial vessels.

Exclusion Criteria:

* Patients with coronary artery disease, hypertensive heart disease, rheumatic valvular heart disease, myocarditis, and other secondary cardiomyopathies.
* poor angiographic image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years with angiography-confirmed absence of coronary stenosis and a definitive diagnosis of dilated cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | At 5-year follow-up
  A composite of cardiac death, hospitalization for heart failure, heart transplantation, and device implantation

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China